CLINICAL TRIAL: NCT07403565
Title: To Evaluate the Efficacy and Safety of the Insulin Patch Pump System in Patients With Diabetes: A Prospective, Randomized, Positive Parallel Controlled, Open-label, Multicenter, Non-inferiority Clinical Trial.
Brief Title: To Evaluate the Efficacy and Safety of the Insulin Patch Pump System in Patients With Diabetes.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suzhou Hechun Medical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20250041-0002
Record Dates: First submitted 2025-12-15; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Type 1 Diabetes; Type 2 Diabetes
Keywords: Non-inferiority; diabetes; insulin patch pump
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (2):
- Insulin Patch Pump System (Experimental): patients who enrolled in this arm use the Insulin Patch Pump System
  Interventions: Device: Insulin Patch Pump System
- Minimed 700 (Active Comparator): patients who enrolled in this group use Minimed 700
  Interventions: Device: Minimed 700

INTERVENTIONS:
Device: Insulin Patch Pump System — patients who enrolled in this group use the Insulin Patch Pump System
  Arms: Insulin Patch Pump System
Device: Minimed 700 — patients who enrolled in this group use Minimed 700
  Arms: Minimed 700

SUMMARY:
Patients will be enrolled and randomly assigned to either the test group or the control group for short-time intensive insulin therapy in inpatient setting. The test group will receive treatment with the Insulin Patch Pump System, while the control group will be treated with the Medtronic MMT-1805 insulin pump (MiniMed 700). The treatment period will last 7 days, during which blood glucose monitoring will be conducted in both groups.

DETAILED DESCRIPTION:
The efficacy and safety of the Insulin Patch Pump System for insulin infusion therapy in patients with diabetes are evaluated by comparing it with the MMT-1805 insulin pump (MiniMed 700). This clinical trial employs a prospective, randomized, active-controlled, open-label, multicenter, non-inferiority design.

On Day 0 (baseline), all participants maintain their pre-existing antidiabetic regimens to collect baseline glucose data. From Day 1 to Day 7, patients undergo a 7-day course of intensive insulin pump therapy. The test group receives treatment with the Insulin Patch Pump System, while the control group is treated with the Medtronic MMT-1805 insulin pump (MiniMed 700). During the intervention, participants receive standardized diabetic hospital meals and perform eight-point daily capillary blood glucose (BG) monitoring. Concurrently, continuous glucose monitoring (CGM) is maintained. Glycated albumin (GA) levels are assessed at baseline (Day 0) and post-treatment (Day 8).

ELIGIBILITY:
Inclusion Criteria:

1. Age is ≥18 years and ≤ 75 years old, gender not restricted;
2. Body Mass Index (BMI) < 30 kg/m²;
3. Patients diagnosed as type 1 diabetes or type 2 diabetes according to WHO standards (1999), and requiring intensive insulin therapy;
4. HbA1c > 7.0% and ≤ 12.0%.

Exclusion Criteria:

1. Those who had used any of the following insulin secretagogues or incretin drugs 14 days prior to enrollment, including sulfonylurea drugs, glinide drugs, dipeptidyl peptidase IV inhibitors (DPP-4i), and glucagon-like peptide-1 receptor agonists (GLP-1RA), among which the weekly formulation of exenatide for GLP-1RA needs to be extended to 70 days prior to enrollment;
2. Pregnant or lactating women;
3. Patients with acute metabolic complications of diabetes (such as diabetic ketoacidosis, non-ketotic hyperosmolar coma, lactic acidosis, etc.) or with hyperglycemia who are receiving intravenous antibiotic treatment due to infection;
4. Within the 28 days prior to enrollment, there was a history of a severe hypoglycemic event (Grade 3 hypoglycemia: without a specific blood glucose threshold, involving severe events with changes in consciousness and/or physical condition, requiring assistance from others);
5. Include patients with other endocrine disorders that may cause abnormal blood sugar levels, such as Cushing's syndrome, primary aldosteronism, and endocrine gland tumors;
6. Patients with acute-stage cardiovascular and cerebrovascular diseases;
7. Patients with a history of allergy to insulin, insulin pump adhesives, or subcutaneous infusion tubes;
8. For patients whose researchers have determined that there are adverse conditions in the skin area where the insulin pump is implanted (such as subcutaneous nodules, subcutaneous fat hyperplasia, subcutaneous fat atrophy, skin scarring, skin infection, skin edema, etc.) that affect the injection and absorption of the medication;
9. Within 14 days prior to enrollment, and during the trial period, the participant had used and planned to use systemic glucocorticoids (excluding inhalation, topical eye medication, or local application);
10. During the screening process, the laboratory test indicators must meet the following criteria: ① Liver function impairment: ALT or AST is greater than 3 times the upper limit of the normal value; ② Kidney function impairment: Serum creatinine is greater than 1.5 times the upper limit of the normal value.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2025-06-14 (Actual); Primary Completion 2025-11-08 (Actual); Study Completion 2025-12-03 (Actual)

PRIMARY OUTCOMES:
Change in mean blood glucose from baseline(Day 0) to Day 7 | Compare the difference in the change of mean blood glucose from baseline (Day 0) to Day 7 between the two groups

SECONDARY OUTCOMES:
Change in mean preprandial blood glucose from baseline(Day 0) to Day 7 | Compare the difference in the change of mean preprandial blood glucose from baseline (Day 0) to Day 7 between the two groups
Change in mean 2-hour postprandial blood glucose from baseline(Day 0) to Day 7 | Compare the difference in the change of mean 2-hour postprandial blood glucose from baseline (Day 0) to Day 7 between the two groups
Change in postprandial glucose excursion (PPGE) from baseline(Day 0) to Day 7 | Compare the difference in the change of postprandial glucose excursion (PPGE) from baseline (Day 0) to Day 7 between the two groups.
Time in Range (TIR) during the treatment period | Compare the difference in TIR between the two groups during the treatment period (Day 1 to Day 7).
Glucose coefficient of variation during the treatment period | Compare the difference in glucose coefficient of variation between the two groups during the treatment period (Day 1 to Day 7).
Change in glycated albumin (GA) | Compare the difference in changes in glycated albumin (GA) between the two groups from Day 0 to Day 8
Time Above Range (TAR) during the treatment period | Compare the difference in TAR between the two groups during the treatment period (Day 1 to Day 7)
Time Below Range (TBR) during the treatment period | Compare the difference in TBR between the two groups during the treatment period (Day 1 to Day 7)
Incidence of diabetic ketoacidosis (DKA) during the treatment period | Day 0 to Day 7
Device defect rate during the treatment period | Day 1 to Day 7
Local injection site reactions during the treatment period | Day 1 to Day 7
Occurrence of adverse events during the treatment period | Day 0 to Day 7
Device performance assessment scale | Day 8
  After completing the training, the investigators administered treatment using the device in accordance with the Instructions for Use. Upon completion of treatment, the investigators rated the device's performance across 11 dimensions, including Ease of device assembly/Ease of parameter configuration/Ease of consumable replacement/Product sealing integrity/Infusion smoothness/Adhesion stability/Battery life/Alarm reliability/Failure-free operation/User interface smoothness/Bluetooth Function and Connection Stability. Each item was scored on a 3-point scale (3 = excellent, 2 = satisfactory, 1 = poor), with higher scores indicating better performance.
Patient satisfaction assessment scale | Day 8
  After treatment completion, subjects rated their satisfaction with the device's ease of use and operation across 5 dimensions, including Implantation Pain Satisfaction/Comfortable Satisfaction/Convenient Satisfaction/Blood Glucose Management Satisfaction/Treatment Satisfaction. Each item was scored on a 3-point scale (3 = excellent, 2 = satisfactory, 1 = poor), with higher scores indicating a more favorable outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohui Guo, Doctor, Principal Investigator — Peking University First Hospital; Zhifeng Cheng, Doctor, Principal Investigator — The Fourth Hospital of Harbin Medical University; Meng Ren, Doctor, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University; Qi Xu, Doctor, Principal Investigator — Second Affiliated Hospital of Shantou University Medical College; Yu Liu, Doctor, Principal Investigator — Nanjing Medical University
Locations (5):
- China (5):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Sun Yat-sen Memorial Hosipital,Sun Yat-sen University, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Shantou University Medical College, Shantou, Guangdong
  - The Fourth Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Sir Run Run Hospital, Nanjing Medical University, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: No